CLINICAL TRIAL: NCT00180674
Title: Anticoagulation for Liver Fibrosis in Patients With Hepatitis C Virus Infection: Pilot Study
Brief Title: Anticoagulation in Liver Fibrosis in Patients With Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: aclf01
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Liver Fibrosis
Keywords: Hepatic fibrosis; anticoagulation; Coumarin; Warfarin; Chronic hepatitis C virus infection
MeSH Terms: conditions — Liver Cirrhosis | interventions — Warfarin

STUDY DESIGN:
Intervention Model Description: The study employed a single centred, prospective, open labelled design. Practical as well as safety concerns dictated that the study could not be conducted in a blinded fashion, since patients taking anticoagulation require monitoring. The study consisted of two 8 week phases: Phase 1 and Phase 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Warfarin anticoagulation (Experimental): Anticoagulated with warfarin to maintain an INR of 2-3 between 8 and 16 weeks (treatment period).
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin

SUMMARY:
Patients who have been treated for hepatitis C virus (HCV) infection who have failed to respond to anti-viral treatment are often concerned about their ongoing liver disease and are therefore looking for alternative treatments which might prevent fibrosis progression. This view is endorsed by patient representative groups (including Charles Gore at the HepC Trust) who have welcomed this trial protocol.

The study is a single centred, prospective, open labelled design. Practical as well as safety concerns dictated that the study could not be conducted in a blinded fashion, since patients taking anticoagulation require monitoring. The study consisted of two 8 week phases: Phase 1 and Phase 2. Phase 1 (observation phase, 0 to 8 weeks) and Phase 2 (treatment phase with warfarin anticoagulation, 8 to 16 weeks). Study completed at end of Phase 2.

DETAILED DESCRIPTION:
Background:

Convincing evidence exists outlining a role for the coagulation system in the pathogenesis of liver fibrosis. In vivo and in vitro studies have suggested a role for thrombin and FXa in activating hepatic stellate cells and epidemiological studies have demonstrated that prothrombotic states accelerate liver fibrosis (Wright et al., 2003).

Hence if prothrombotic states accelerate liver fibrosis, conversely anticoagulation should slow liver fibrosis. Animal studies have confirmed this (Anstee et al., 2008; Duplantier et al., 2004), and confirmed the beneficial effect of inhibiting the coagulation cascade. The number of patients with HCV infection on anticoagulants is small and there is no published case series. Similarly there are problems assessing disease progression using patients with haemophilia and HCV infection. The therapeutic use of anticoagulation to prevent fibrosis in humans is not without precedent, and warfarin has demonstrated a survival benefit in pulmonary fibrosis (Kubo et al., 2005).

The antifibrotic potential of warfarin anticoagulation needs to be formally assessed in the setting of a clinical trial using patients with documented liver fibrosis. Most previous human studies of antifibrotics have taken place in patients with chronic HCV infection who have failed anti-viral therapy, as they are a model of progressive fibrosis (Anstee et al., 2009).

Study aims:

1. To evaluate if any potential effect on the progression of liver fibrosis in patients infected with Hepatitis C virus, with moderate severity liver fibrosis is demonstrable with anticoagulation.
2. To evaluate the safety of anticoagulation in patients infected with Hepatitis C virus infection, with moderate severity liver fibrosis.

Patients:

The study was approved by the St. Mary's Hospital Ethics committee and conducted in accordance with the principles of the Declaration of Helsinki. Potential participants were identified via the departmental Hepatitis C database. All potential candidates were screened for the inclusion and exclusion criteria.

Inclusion criteria:

Patients were eligible for inclusion if they were aged greater than 17 years of age, had evidence of active Hepatitis C viral replication (HCV RNA PCR positive), ALT of greater than 40 iu/ml, a modified histology activity index fibrosis score (Ishak et al., 1995) of greater than 2 but less than 5 on liver biopsy within the last five years, and had failed antiviral therapy for Hepatitis C in the last 5 years.

Exclusion criteria:

Patients requiring anticoagulation for existing clinical indications; standard contraindications to anticoagulation (active peptic ulcer disease, past history of haemorrhagic stroke, thrombocytopaenia, platelets count < 100 x109 /L); clinical evidence of portal hypertension; known cerebrovascular abnormalities; HIV antibody positive; alcohol abuse (> 40 units/week); menhorragia and pregnancy.

Potential qualifying subjects were initially contacted by telephone to be informed about the study and arrange a formal screening visit. During the screening visit, entry criteria were confirmed and all patients who agreed to participate were required to give written informed consent.

Study design:

The study employed a single centred, prospective, open labelled design. Practical as well as safety concerns dictated that the study could not be conducted in a blinded fashion, since patients taking anticoagulation require monitoring. The study consisted of two 8 week phases: Phase 1 and Phase 2.

Phase 1 (Week 0 to Week 8) Phase 1 of the study consisted of 8 weeks of observation, which commenced following a baseline visit at week 0. At the baseline study routine blood tests and non-invasive markers of fibrosis were performed. No placebo was given during the observation period. At week 8 patients underwent their second study visit during which routine blood tests and evaluation with non-invasive markers of fibrosis were repeated. The week 8 study visit marked the completion of Phase 1, following which patients entered Phase 2 of the study.

Phase 2 (Week 8 to Week 16) Phase 2 of the study consisted of 8 weeks of anticoagulation with warfarin. In previous animal studies (Anstee et al., 2008), warfarin anticoagulation to achieve a whole blood clotting of twice the normal range was sufficient to retard fibrosis significantly, hence the international normalised ration (INR) was aimed to be maintained between 2 to 3 during the treatment period. Patients were given a standard induction regimen of warfarin in keeping with the outpatient warfarin loading protocol of the hospital's anticoagulation clinic. Warfarin was supplied by the hospital pharmacy. Routine INR monitoring and warfarin dosing was undertaken by the anticoagulation clinic on a weekly basis. Patients were monitored at these visits for any adverse events related to the treatment. At week 16, following 8 weeks of anticoagulation, a further study visit was organised. Routine bloods tests and non-invasive markers of fibrosis were performed at this visit, which marked the completion of each patient's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged >17 years (male and female)
* HCV infection PCR positive
* ALT > 40 iu/ml
* Ishak fibrosis score (within last 5 years) > 2, < 5
* Informed consent
* Failed antiviral therapy for HCV in last 5 years

Exclusion Criteria:

* Patients requiring anticoagulation for existing clinical indications
* Active peptic ulcer disease
* Past history of haemorrhagic stroke
* Thrombocytopaenia (platelets count < 100 x 109 /L)
* Clinical evidence of portal hypertension
* Known cerebrovascular abnormalities;
* HIV antibody positive;
* Alcohol abuse (>40 unites/week)
* Menhorragia
* Pregnancy

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-08; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Thursz, MBBS, FRCP, Principal Investigator — St Mary's Hospital & Imperial College London
Locations (1):
- St Mary's Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Result publication — https://gut.bmj.com/content/59/Suppl_2/A18.2

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14 patients were enrolled in the study. Ten patients completed the study. Four patients withdrew from the study, all during the Phase 1 Observation Period due to personal reasons. These 4 patients did not participate in Phase 2, Treatment Period and they are not included in the analyses.
Groups:
- Warfarin Anticoagulation: Anticoagulated with warfarin to maintain an INR of 2-3 between 8 and 16 weeks (Phase 2, Treatment Period).
Period: Phase 1, Observation Period
Arm/Group | Warfarin Anticoagulation
Started | 14
Completed | 10
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: Phase 2, Warfarin Treatment Period
Arm/Group | Warfarin Anticoagulation
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Warfarin Anticoagulation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 49.5 [42 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Median Liver Stiffness Value
Description: Median liver stiffness at 16-weeks following the 8-week period of anticoagulation, compared to 8-week period of observation.
  kPa values reported are the values from completion of the period of anticoagulation at week 16 versus completion of the observation period at week 8, and start of the observation period at week 0.
Time Frame: Baseline (start of the observation period at week 0), 8-weeks (completion of the observation period) and 16-weeks (completion of the period of anticoagulation)
Population: One participant excluded from Phase 2, Warfarin Anticoagulation Period due to a non serious adverse event.
Measure: Median (Inter-Quartile Range); unit: kPa
Groups:
- Observation Period: Phase 1, Observation Period Observation period began at Week 0 and was completed at Week 8.
- Warfarin Anticoagulation: Phase 2, Treatment Period Anticoagulated with warfarin to maintain an INR of 2-3 between 8 and 16 weeks (treatment period).
Arm/Group | Observation Period | Warfarin Anticoagulation
Number analyzed (Participants) | 10 | 9
kPa | 7.70 [NA to NA] — The PI has left the institution and we have exhausted all efforts to locate this data. No data is available and therefore cannot be reported. | 6.90 [NA to NA] — The PI has left the institution and we have exhausted all efforts to locate this data. No data is available and therefore cannot be reported.
Statistical Analysis 1: Comparison: Observation Period; Test type: Superiority; p = 0.043, Wilcoxon Signed Ranks test

2. Secondary Outcome: Number of Participants With Adverse Events
Description: The secondary endpoints were the proportion of patients with a reduction in serum markers of fibrosis and HTTs following the 8-week period of anticoagulation compared to the 8-week period of observation and the safety of anticoagulation defined by the number of adverse events.
Time Frame: 8-week period of warfarin treatment and 8-week observation period (16 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Observation Period: Phase 1, Observation Period Phase 1 of the study consisted of 8 weeks of observation, which commenced following a baseline visit at week 0.
- Warfarin Treatment Period: Phase 2, Treatment Period:
  Anticoagulated with warfarin to maintain an INR of 2-3 between 8 and 16 weeks (treatment period).
Arm/Group | Observation Period | Warfarin Treatment Period
Number analyzed (Participants) | 10 | 9
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Observation Period (Phase 1): Phase 1, Observation Period Phase 1 of the study consisted of 8 weeks of observation, which commenced following a baseline visit at week 0.
- Warfarin Anticoagulation (Phase 2: Phase 2, Treatment Period Anticoagulated with warfarin to maintain an INR of 2-3 between 8 and 16 weeks (treatment period).
  A single adverse event was noted in one subject during the anticoagulation period. This was classed as minor in severity and related to an episode of minor haemorrhage secondary to an episode of gingivitis, which resolved following antibiotics and did not require blood transfusion, but did require cessation of the anticoagulation for a short period of 2 days. This patient was not included in the analysis. No other subjects required cessation of treatment during the anticoagulation period.
Arm/Group | Observation Period (Phase 1) | Warfarin Anticoagulation (Phase 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation Period (Phase 1) (N=10) | Warfarin Anticoagulation (Phase 2 (N=9)
Minor haemorrhage (General disorders) | 0 (0) | 1 (1) — An episode of minor haemorrhage secondary to an episode of gingivitis, which resolved following antibiotics and did not require blood transfusion, but did require cessation of the anticoagulation for a short period of 2 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes